CLINICAL TRIAL: NCT03424525
Title: 11C-Trimethoprim PET/CT Imaging to Evaluate Biodistribution and Kinetics in Human
Brief Title: 11C-Trimethoprim PET/CT Imaging to Evaluate Biodistribution and Kinetics in Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, David Mankoff, Principal Investigator, University of Pennsylvania
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 827333
Record Dates: First submitted 2017-12-07; First posted 2018-02-07 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Biodistribution (Experimental): The Biodistribution cohort referred from orthopedics who will undergo a series of vertex to mid-thigh (or feet if indicated) biodistribution [11C]trimethoprim PET/CT scans over a period of approximately 2 ½ hours.
  Interventions: Drug: 11C-Trimethoprim
- Dynamic (Experimental): The Dynamic cohort will undergo approximately 60 minutes of dynamic scanning followed by up to 2 static skull base to mid-thigh (or feet if indicated) scans imaging post injection of [11C]trimethoprim. Some subjects who may be selected clinically to undergo surgical or antibiotic treatment may undergo a second therapy may also undergo an optional second [11C]trimethoprim PET/CT after the initiation of therapy to collect pilot data on the changes in [11C]trimethoprim biodistribution and uptake with therapy, the timing of this scan may vary depending on the type of treatment the patient is receiving.
  Interventions: Drug: 11C-Trimethoprim

INTERVENTIONS:
Drug: 11C-Trimethoprim — [11C]TMP is a radiolabeled imaging agent for positron emission tomography (PET/CT). Most relevant to this protocol, it is for imaging bacterial infection in human subjects. TMP is well-known, safe, broad-spectrum, synthetic, small molecule antibiotic that has been used clinically for over 50 years for the treatment of acute bacterial infection and has been combined with sulfa-based antibiotics (Bactrim/Septra) for bacterial infection prophylaxis especially in the lung and bladder.

SUMMARY:
Patients with suspected bacterial infection at the time screening are eligible for this study. Patients may participate in this study if they are at least 18 years of age, and most participants will be receiving care at the clinical practices of the University of Pennsylvania. Up to 30 subjects will participate in two different imaging cohorts.

The Biodistribution cohort will include up to 5 patients referred from orthopedics who will undergo a series of vertex to mid-thigh (or feet if indicated) biodistribution [11C]trimethoprim PET/CT scans over a period of approximately 2 ½ hours.

The Dynamic cohort will include up to 25 patients who will undergo approximately 60 minutes of dynamic scanning followed by up to 2 static skull base to mid-thigh (or feet if indicated) scans imaging post injection of [11C]trimethoprim. Some subjects who may be selected clinically to undergo surgical or antibiotic treatment may undergo a second therapy may also undergo an optional second [11C]trimethoprim PET/CT after the initiation of therapy to collect pilot data on the changes in [11C]trimethoprim biodistribution and uptake with therapy, the timing of this scan may vary depending on the type of treatment the patient is receiving.

Patients will also undergo baseline lab tests complete blood count (CBC), C-reactive protein (CRP), erythrocyte sedimentation rate (ESR) and blood cultures. If these tests are done as part of clinical standard of care they will not need to be repeated for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion Criteria at least 18 years of age
2. Known or suspected bacterial infection.
3. Participants must be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria:

1. Antibiotic therapy with trimethoprim within 48h of the baseline PET/CT scan.
2. Inability to tolerate imaging procedures in the opinion of an investigator or treating physician
3. Serious or unstable medical or psychological comorbidities that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study.
4. Females who are pregnant or breast feeding at the time of screening will not be eligible for this study; a urine pregnancy test will be performed in women of child-bearing potential at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Kinetics of uptake of [11C]TMP in human patients | 3 years
  The biodistribution which includes kinetics of uptake of [11C]TMP in human patients via PET/CT will be measured

SECONDARY OUTCOMES:
[11C]trimethoprim in infected versus non-infected tissues | 3 years
  Measure uptake of [11C]trimethoprim in infected versus non-infected tissues via PET/CT
The change in biodistribution which includes kinetics of uptake of [11C]TMP in human patients after therapy | 3 years
  Describe the change in biodistribution which incldues kinetics of uptake of [11C]TMP in human via PET/CT

CONTACTS AND LOCATIONS:
Overall Officials: David Mankoff, MD PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Young AJ, Doot RK, Cho JK, Pham JM, Ordonez AA, Del Castillo AF, Dominguez TL, Dugyala S, Schubert EK, Lee H, Pantel AR, Mach RH, Mankoff DA, Sellmyer MA. First-in-Human Biodistribution and Dosimetry of [11C]Trimethoprim. Mol Imaging Biol. 2025 Nov 22. doi: 10.1007/s11307-025-02064-7. Online ahead of print. PMID 41275068
- [Derived] Lee IK, Jacome DA, Cho JK, Tu V, Young AJ, Dominguez T, Northrup JD, Etersque JM, Lee HS, Ruff A, Aklilu O, Bittinger K, Glaser LJ, Dorgan D, Hadjiliadis D, Kohli RM, Mach RH, Mankoff DA, Doot RK, Sellmyer MA. Imaging sensitive and drug-resistant bacterial infection with [11C]-trimethoprim. J Clin Invest. 2022 Sep 15;132(18):e156679. doi: 10.1172/JCI156679. PMID 36106638